CLINICAL TRIAL: NCT04723108
Title: Virtual Reality as a Symptom Control Intervention for Women With Gynecologic Cancer Receiving Chemotherapy: A Pilot Proof of Concept Study
Brief Title: Virtual Reality for Chemotherapy Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment and researcher left the institution
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAS5430
Record Dates: First submitted 2021-01-22; First posted 2021-01-25 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Oncologic Complications
Keywords: chemotherapy; side effects; gynecologic cancers; meditative experience; virtual reality (VR)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Virtual reality arm (Experimental): Participants will be asked to use virtual reality during their infusion for a duration of at least 10 minutes.
  Interventions: Other: Destek V4 Virtual Reality Headset

INTERVENTIONS:
Other: Destek V4 Virtual Reality Headset — The DESTEK V4 is a smartphone VR headset made by DESTEK, a manufacturer based in the US. This mobile virtual reality headset is compatible with most iOS and Android smartphones, as long as their screen size is between 4.5 and 6.

SUMMARY:
The purpose of this feasibility prospective study is to explore if the use of virtual reality as a distraction intervention for women with gynecologic cancer during chemotherapy administration reduces adverse symptoms. In this study, the treatment participants serve as their own control. The study will be performed over a 3 month period limit in order to assess implementation capability and symptom management of gynecologic cancer patients receiving chemotherapy treatment at Columbia University Irving Medical Center (CUIMC).

DETAILED DESCRIPTION:
Gynecologic cancer encompasses various conditions such as uterine, ovarian, cervical, peritoneal, fallopian tube, vaginal and vulvar cancers. Of these, uterine cancer is the top 4th cancer diagnosed and ovarian cancer the 5th deadliest in women.

Many of these patients require some form of chemotherapy administration during their treatment course. Chemotherapy is given at different stages of the treatment course with some patients receiving it prior to surgical intervention (neo-adjuvant), post-surgical intervention (adjuvant), and in the recurrent disease setting. Chemotherapy infusions can cause distressing side effects to the patients in the form of physical and also emotional/psychological effects, which may disrupt compliance to treatment protocols. Physical symptoms often begin during the administration of chemotherapy, such as nausea, vomiting, fatigue, pain, and anorexia. As a result, patients frequently experience psychological distress, including feelings of depression, helplessness, anxiety, and cognitive decline. These directly interfere with the patient's ability to perform activities of daily living and daily quality of life. The purpose of this study is to assess the effect of virtual reality (VR) sessions as a distraction intervention at time of chemotherapy infusion on symptom control.

VR creates an alternative, 'less stressful' environment, and is easy to use. Users of VR wear a head-mounted display with a close proximity screen that creates a sense of being transported into a 3-dimensional world. The technology can be individualized to be interactive, and allows for an immersion experience by engaging several senses simultaneously. Importantly, VR has become increasingly portable, immersive and inexpensive to adopt. VR does not require a subject's experience or competency prior to use in the clinical setting. VR has been used to assess and treat a wide variety of medical, surgical, psychiatric, and neurocognitive conditions including pain, addiction, anxiety disorders, schizophrenia, eating disorders, and stroke rehabilitation.

There have also been functional MRI studies demonstrating the effect of VR on the brain during receipt of painful stimuli. Multiple studies have demonstrated the benefit of VR as a distraction intervention for decreasing symptom distress, particularly in regards to anxiety, distress and fatigue, and have demonstrated that it is feasible to integrate in the chemotherapy setting for patients receiving treatments for various cancers, as well as when enduring medical procedures.

In summary, VR has been shown to be safe and effective in reducing emotional distress of patients undergoing chemotherapy. These studies are generally limited in small sample size, but all have shown to be safe and feasible. To date, the benefit of VR during chemotherapy infusion has not been evaluated in patients with gynecologic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. All gynecologic oncology patients undergoing intravenous (IV) chemotherapy as standard of care treatment for their disease.
2. Age greater than or equal to 18 years
3. Patients willing to participate on surveys prior to and post chemotherapy infusion treatments
4. Patient must own or have access to an iphone or android device with virtual reality application capability

Exclusion Criteria:

1. Patients with hearing impairment
2. Patients with known balance disorders such as vertigo/cybersickness
3. Patients with known history of epileptic seizures
4. Patients who are unable to wear the virtual reality headset
5. Patients who are not receiving pre-chemotherapy labs as part of their standard treatment protocol
6. Patients who receive additional intravenous medications, such as antihypertensives, steroids, analgesics, anxiolytics during chemotherapy session that is not part of the standard chemotherapy regimen.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-08-17 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
Symptom Survey A | upto 3 months
  Symptom Survey A will be administered prior to first three chemotherapy infusions. Descriptive statistics will be utilized to characterize the survey question response proportions (i.e., distribution of responses to questions on the survey) (frequency, percent). Estimated differences in survey responses between 1) patient's perception pre-intervention vs. 2) patient's perception post-intervention, will be evaluated by the two-sample t-test, Wilcoxon rank-sum test, chi-square test, and Fisher's exact test, as appropriate. All analyses will be performed in SAS version 9.3
Symptom Survey B | 3-4 months
  Symptom Survey B will be administered after the third chemotherapy infusion. Descriptive statistics will be utilized to characterize the survey question response proportions (i.e., distribution of responses to questions on the survey) (frequency, percent). Estimated differences in survey responses between 1) patient's perception pre-intervention vs. 2) patient's perception post-intervention, will be evaluated by the two-sample t-test, Wilcoxon rank-sum test, chi-square test, and Fisher's exact test, as appropriate. All analyses will be performed in SAS version 9.3

CONTACTS AND LOCATIONS:
Overall Officials: June Y. Hou, MD, Principal Investigator — Columbia University

IPD SHARING:
Plan to Share IPD: No